CLINICAL TRIAL: NCT04840082
Title: Optimal Insertion Length for Nasal Mid-turbinate and Nasopharyngeal Swabs for Respiratory Virus Infection Diagnostic Testing - a Clinical Trial
Brief Title: Optimal Length for Nasal Mid-turbinate and Nasopharyngeal Swabs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tobias Todsen, MD, PhD, Ass. Prof, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21015626
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collecting of Clinical Specimens for COVID-19 Testing (Experimental): Nasopharyngeal swab is performed on all participants to collect specimens for Rapid antigen COVID-19 Testing
  Interventions: Diagnostic Test: Nasopharyngeal swab for COVID-19 testing

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab for COVID-19 testing — A nasopharyngeal swab was performed endoscopically video guided to measure the actual length from to the mid turbinate and the posterior nasopharyngeal wall

SUMMARY:
This study aim to explore the optimal swap insertion length for mid-turbinate and nasopharyngeal samples. Our clinical trial took place at a Covid-19 test center in Copenhagen. Participants consisted of voluntary citizens who were at the test center for a nasopharyngeal antigen quicktest. An endoscopic examination was performed simultaneous with the swap to measure the length from the vestibulum nasi to the posterior wall of the nasopharynx and the mid-turbinate.

ELIGIBILITY:
Inclusion Criteria:

* Referred for COVID-19 testing

Exclusion Criteria:

* Nose patology

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Length from the vestibulum nasi to the posterior wall of the nasopharynx. | From inclusion at the testcenter until the COVID-19 testing was completed.
  Endoscopic measurement of the length from the vestibulum nasi to the posterior wall of the nasopharynx.
Length from the vestibulum nasi to the mid-turbinate. | From inclusion at the testcenter until the endoscopic examination was completed
  Endoscopic measurement of the length from the vestibulum nasi to the mid-turbinate.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen East, Denmark

IPD SHARING:
Plan to Share IPD: Undecided